CLINICAL TRIAL: NCT01119053
Title: Effects of Vagus Nerve Stimulation (VNS) as a Treatment of Persistent Depression With Comorbid Personality Disorders (Impulse-VNS
Acronym: Impuls-V
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Claus Wolff-Menzler, Dr, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01VNS2009
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Depression; Comorbid Personality Disorders
Keywords: VNS; Depression; Personality-Disorder; Stimulation
MeSH Terms: conditions — Depression; Personality Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Sham Comparator): In this branch of study, study participants obtain the VNS therapy after a defined space of time of 12 weeks.
  Interventions: Device: VNS Pulse Model 102
- Arm II (Experimental): Within this space of time, study participants obtain the VNS therapy at once.
  Interventions: Device: VNS Pulse Model 102

INTERVENTIONS:
Device: VNS Pulse Model 102 — Individual dosage within the realm of 0,25 mA - 3,5 mA. Uninterrupted stimulation of 24 h.
  Arms: Arm II
Device: VNS Pulse Model 102 — Within this branch, study participants obtain the VNS therapy after a defined space of time of 12 weeks.
  Arms: Arm I

SUMMARY:
In this monocentre two-armed double blind randomised placebo-controlled study - in which the control group obtains the VNS therapy within a defined space of time after 12 weeks - the impact of vagus nerve stimulation on depressive symptomatology of patients with therapy-resistant depressive personality disorders shall be analysed. Particularly in comorbid disorders, medicamentous treatment shows exceedingly bad response rates. Against the background of hitherto insufficient treatment strategies for chronic or persistent depression with comorbidities, the proceeding of a study on the effects of VNS on depressive patients with comorbid disorders is absolutely essential.

ELIGIBILITY:
Inclusion criteria

* embedding criteria according to "VNS manual for doctors"
* diagnosis of a recurrent depressive disorder (based on ICD-10 criteria) and a comorbid personality disorder (according to SKID I/II) with an ailment period of more than six months
* age 18-80 years
* verbal IQ (WST) 85 points
* HAM-D sum score > 20 points
* at least four depressive episodes in the anamnesis
* no amelioration of current depressive episodes under two different antidepressants in appropriate dosage for six weeks
* constant medication within the last two weeks (at the discretion of the supervising doctor)
* written consent after informing the patient about the study
* no VNS treatment to date
* no misuse of illegal drugs or alcohol
* Women in childbearing age are not permitted to participate in the study if a doctor has asserted the non-existence of pregnancy before the beginning of the study. Furthermore, the procedure of a pregnancy test is recommended after the completion of the study. During the study, a reliable type of contraception (such as the Pill) should be taken. The doctor provides further information.

Exclusion criteria according to "VNS manual for the doctor"

* present hospitalisation according to the federal states' PsychKG
* clinically relevant unstable bodily concomitant diseases
* former VNS treatment
* reduction of intelligence with verbal IQ < 85 (WST)
* conceivable use of an MRT examination after the implantation of the VNS-system
* for diagnostic examinations with the dTMS and the MRT: electric devices (such as cardiac pacemakers, medicine pumps etc.) or pieces of metal (ferromagnetic, e.g. screws after bone fractures) within or at the body, or large-scale tattoos
* conditions that do not allow to use VNS, such as relevant dysfunctions of the heart's stimulus conduction system or cardiac arrhythmia, stomach ulcer, dysphagia, palsy of parts of the n-vagus nerve
* insufficient knowledge of the German language
* pregnancy or lactation
* current misuse of substances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
To analyse whether VNS is effective within the therapy of depression with comorbid personality disorders | 6 Month
  The primary objective of this study is to analyse whether VNS is effective within the therapy of depression with comorbid personality disorders.
  It shall be verified, as a primary hypothesis, whether VNS with ongoing stimulation is significantly predominant to a non-stimulating control with respect to reducing depressive symptomatology (for differences within HAM-D score and the response rate as the percentage of patients with a reduction in the HAM-D score of at least 50%, week 1 - week 12, see flow-chart).

SECONDARY OUTCOMES:
Acquisition of Alteration by means of BDI, TMT-A and B, WMS R, VLMT; WHO-QoL, GAF, CGM, SDS | 6 month
  Acquisition of the improvement of self-rated depressiveness (BDI), stress axis (cortisol of neurocognition, quality of life (WHO-QoL) and impairment through disease (GAF, CGI, SDS), examination of brain structural and functional parametres as predictors for therapy response (VBM-MRT), Region of Interest Approach and proton magnetic resonance spectroscopy, diagnostic TMS (dTMS) in the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Falkai, MD, Study Director — Dept. of Psychiatry and Psychotherapy (University Medical Centre Goettingen, Germany); Claus Wolff-Menzler, MD, Principal Investigator — Dept. of Psychiatry and Psychotherapy (University Medical Centre Goettingen, Germany)
Locations (1):
- Dept. of Psychiatry and Psychotherapy (University Medical Centre), Göttingen, Lower Saxony, Germany

REFERENCES:
- See also: Dept. of Psychiatry and Psychotherapy (University Medical Centre Goettingen) — http://www.psychiatrie.med.uni-goettingen.de/